CLINICAL TRIAL: NCT00012259
Title: A Phase II Study Of Troxatyl In Patients With CML Blastic Phase Disease
Brief Title: Troxacitabine in Treating Patients With Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCH-4556-214; CDR0000068498 (Registry Identifier: PDQ (Physician Data Query)); NCI-V01-1648
Record Dates: First submitted 2001-03-03; First posted 2004-02-26 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Leukemia
Keywords: relapsing chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; chronic myelogenous leukemia, BCR-ABL1 positive
MeSH Terms: conditions — Leukemia; Blast Crisis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — troxacitabine

ARMS (1):
- troxacitabine (Experimental)
  Interventions: Drug: troxacitabine

INTERVENTIONS:
Drug: troxacitabine
  Other Names: 8 mg/m2 administered IV over 30 minutes per day for 5 consecutive days

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of troxacitabine in treating patients who have blast phase chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate, in terms of achieving complete hematologic remission, partial hematologic remission, hematologic improvement, partial response, or back to chronic phase status, in patients with blastic phase chronic myelogenous leukemia treated with troxacitabine. II. Determine the proportion of patients whose disease returns to chronic phase and remains at that level for at least 3 months when treated with this drug. III. Determine the toxicity profile of this drug in these patients. IV. Determine the duration of survival of patients treated with this drug.

OUTLINE: This is a multicenter study. Patients receive troxacitabine IV over 30 minutes on days 1-5. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity. Patients are followed every 4 weeks until relapse.

PROJECTED ACCRUAL: A maximum of 50 patients will be accrued for this study within 14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of Philadelphia chromosome-positive blastic phase chronic myelogenous leukemia (CML) with blasts of non-lymphoid origin Blastic phase defined as: At least 30% blasts in the blood or bone marrow OR Presence of extramedullary infiltration outside the liver or spleen No leukemic CNS involvement

PATIENT CHARACTERISTICS: Age: 16 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2.0 mg/dL AST or ALT less than 3 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine less than 1.8 mg/dL if creatinine clearance at least 45 mL/min Other: No known hypersensitivity to troxacitabine or its analogues No active uncontrolled serious infection No other severe medical condition that would preclude study No neurologic or psychiatric disorders that would preclude informed consent No uncontrolled underlying medical condition or underlying condition that could be aggrevated by treatment Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 24 hours since prior hydroxyurea Prior STI571 for blastic phase chronic myelogenous leukemia allowed No other prior chemotherapy for blastic phase disease Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified Other: At least 14 days since prior investigational agents and recovered No other concurrent investigational agents

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2000-12-11 (Actual); Primary Completion 2002-03-27 (Actual); Study Completion 2002-03-27 (Actual)

PRIMARY OUTCOMES:
Conventional Response Rate | Week 4
  Conventional Response Rate defined as the achievement of complete hematologic remission (CHR), partial hematologic remission (PHR), hematologic improvement (HI), partial response (PR), or back to chronic phase (BCP).
Conventional Response Rate | Week 8
  Conventional Response Rate defined as the achievement of complete hematologic remission (CHR), partial hematologic remission (PHR), hematologic improvement (HI), partial response (PR), or back to chronic phase (BCP).
Conventional Response Rate | Week 12
  Conventional Response Rate defined as the achievement of complete hematologic remission (CHR), partial hematologic remission (PHR), hematologic improvement (HI), partial response (PR), or back to chronic phase (BCP).
Conventional Response Rate | Week 16
  Conventional Response Rate defined as the achievement of complete hematologic remission (CHR), partial hematologic remission (PHR), hematologic improvement (HI), partial response (PR), or back to chronic phase (BCP).
Conventional Response Rate | Week 20
  Conventional Response Rate defined as the achievement of complete hematologic remission (CHR), partial hematologic remission (PHR), hematologic improvement (HI), partial response (PR), or back to chronic phase (BCP).
Conventional Response Rate | Week 24
  Conventional Response Rate defined as the achievement of complete hematologic remission (CHR), partial hematologic remission (PHR), hematologic improvement (HI), partial response (PR), or back to chronic phase (BCP).
Conventional Response Rate | Week 28
  Conventional Response Rate defined as the achievement of complete hematologic remission (CHR), partial hematologic remission (PHR), hematologic improvement (HI), partial response (PR), or back to chronic phase (BCP).
Conventional Response Rate | Week 32
  Conventional Response Rate defined as the achievement of complete hematologic remission (CHR), partial hematologic remission (PHR), hematologic improvement (HI), partial response (PR), or back to chronic phase (BCP).
Conventional Response Rate | Week 36
  Conventional Response Rate defined as the achievement of complete hematologic remission (CHR), partial hematologic remission (PHR), hematologic improvement (HI), partial response (PR), or back to chronic phase (BCP).
Conventional Response Rate | Week 40
  Conventional Response Rate defined as the achievement of complete hematologic remission (CHR), partial hematologic remission (PHR), hematologic improvement (HI), partial response (PR), or back to chronic phase (BCP).
Conventional Response Rate | Week 44
  Conventional Response Rate defined as the achievement of complete hematologic remission (CHR), partial hematologic remission (PHR), hematologic improvement (HI), partial response (PR), or back to chronic phase (BCP).
Conventional Response Rate | Week 48
  Conventional Response Rate defined as the achievement of complete hematologic remission (CHR), partial hematologic remission (PHR), hematologic improvement (HI), partial response (PR), or back to chronic phase (BCP).
Conventional Response Rate | Week 52
  Conventional Response Rate defined as the achievement of complete hematologic remission (CHR), partial hematologic remission (PHR), hematologic improvement (HI), partial response (PR), or back to chronic phase (BCP).
Conventional Response Rate | Week 56
  Conventional Response Rate defined as the achievement of complete hematologic remission (CHR), partial hematologic remission (PHR), hematologic improvement (HI), partial response (PR), or back to chronic phase (BCP).
Conventional Response Rate | Week 60
  Conventional Response Rate defined as the achievement of complete hematologic remission (CHR), partial hematologic remission (PHR), hematologic improvement (HI), partial response (PR), or back to chronic phase (BCP).
Conventional Response Rate | Week 64
  Conventional Response Rate defined as the achievement of complete hematologic remission (CHR), partial hematologic remission (PHR), hematologic improvement (HI), partial response (PR), or back to chronic phase (BCP).

SECONDARY OUTCOMES:
Percent of Patients Returning to Chronic Phase | Throughout the study period of approximately 15 months.
Toxicity Profile | Every 4 weeks throughout the study period of approximately 15 months.
Survival Duration | Throughout the study period of approximately 15 months.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (20):
- United States (15):
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Cedars-Sinai Comprehensive Cancer Center, Los Angeles, California
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Northwestern University Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Cancer Center of Albany Medical Center, Albany, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Medical College, Valhalla, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
- Canada (5):
  - Health Sciences Centre, Winnipeg, Manitoba
  - Ottawa General Hospital, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Royal Victoria Hospital - Montreal, Montreal, Quebec